CLINICAL TRIAL: NCT04921579
Title: Evaluation of Treatment Duration of En-masse Versus Two Steps Retraction in Patients Having Maxillary Protrusion: A Randomized Clinical Trial
Brief Title: Evaluation of Treatment Duration of En-masse Versus Two Steps Retraction in Patients Having Maxillary Protrusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Aya Ahmed El Ashwal, principle investigator, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUE.REC (23)/11-2019
Record Dates: First submitted 2021-05-31; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Bimaxillary Protrusion
Keywords: En-masse retraction; two step retraction; friction; retraction time; Dental models

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: single ( Outcomes Assessor) Only the outcome assessors will be blind. The patients name will be sealed from pre and post radiographs and study models. Then two assessors will carry out, blindly and independently, the measurements and analysis of the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- En masse retraction (Experimental): six anterior teeth are retracted by en masse technique using a crimpable hook distal to upper lateral incisor and a power chain.
  Interventions: Procedure: En masse retraction
- two step retraction (Experimental): six anterior teeth are retracted by two step technique by canine retraction followed by four anterior teeth retraction using a crimpable hook distal to upper lateral incisor and a power chain.
  Interventions: Procedure: Two-Step retraction

INTERVENTIONS:
Procedure: En masse retraction — Retraction stated on a 0.017''x 0.025'' Stainless steel wire using elastomeric chain ( force applied 200 g per side) extending between the crimpable hooks and the mini-screw.
  Arms: En masse retraction
Procedure: Two-Step retraction — Retraction of canine started on a 0.017''x0.025'' Stainless steel wire using elastomeric chain ( force applied 150 g per side) followed by anterior teeth retraction on 0.017''x0.025'' Stainless steel wire using elastomeric chain ( force applied 160 g per side) extending between crimpable hooks and the mini-screw.
  Arms: two step retraction

SUMMARY:
Brief summary: there's a scarcity in literature concerning time needed to retract anterior segment following premolars extraction. the purpose of this study is to determine, in orthodontic patients with maxillary protrusion, which form of technique of retraction offers a faster treatment duration of retraction : en-masse or two step techniques

DETAILED DESCRIPTION:
Anterior segment retraction can be done in one of two ways: through En masse or two step techniques. Both are viable options, but, ideally, the investigator wanted to retract and complete the orthodontic treatment as quickly as possible, in order to decrease the negative effects that may occur during treatment. Which of these techniques results in a decreased treatment time is still up for debate.

ELIGIBILITY:
Inclusion Criteria:

* Adults and adolescent patients ( both gender)
* Age range (14- 24)
* patient with maxillary protrusion requiring first premolars extraction ( bimaxillary protrusion or class II division 1 cases)
* patients with fully erupted permanent teeth ( not necessarily including the third molar).
* cases required maximum anchorage during retraction.
* good general and oral health

Exclusion Criteria:

* patients suffering from any systemic diseases interfering with tooth movement.
* patients with extracted or missing permanent teeth (except for third molars).
* patients with badly decayed teeth.
* patients with any parafunctional habits ( i.e. Bruxism, tongue thrusting, mouth breathing, etc.,.....)
* patients with previous orthodontic treatment

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
Time to close extraction space | from pre to post retraction ( an average of 10 - 12 months)
  the antero-posterior movement of anterior teeth are assessed by monthly taken models and patient record sheets

SECONDARY OUTCOMES:
Anchorage loss | From pre to post retraction ( an average of 10- 12 months)
  Digitalized dental models taken before and after completion of retraction will be measured by identifying landmarks and reference lines and planes ( measured in mm)
pain of intervention | From pre to post retraction ( an average of 10 - 12 months)
  Each patient was informed to fill a questionnaire regarding treatment experience in Visual analogue scale scoring from (0 -10) 0 means no pain and 10 means severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Yehia Mostafa, professor and chairman, Study Director — Future University in Egypt
Locations (1):
- Future University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD sharing statement
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after publication

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT04921579/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT04921579/ICF_001.pdf